CLINICAL TRIAL: NCT06901323
Title: Effect of L-carnitine Supplementation on Phenylalanine and Brain-derived Neurotrophic Factor Levels in Infants and Children With Phenylketonuria Two Phases Study 1- Cross Sectional Comparative Study ( PKU Versus Non PKU Infants and Children). 2- Open Label Randomized Controlled Clinical Trial for PKU Patients Only. 1/ Intervention Group: 44 Patients Will Treated With L-carnitine at a Dose of 100 mg/kg/Dose for One Year Beside Their Treatment. 2/ Control PKU Group: 44 Patients Will Not Receive L-carnitine Supplementation Beside Their Treatment 3/ Control Healthy Group Same Age and Sex
Brief Title: Effect of L-carnitine Supplementation on Phenylalanine and Brain-derived Neurotrophic Factor Levels in Infants and Children With Phenylketonuria
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Eman Nabil, Principal Investigator, Mansoura University
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: MD.24.06.860
Record Dates: First submitted 2025-03-24; First posted 2025-03-28 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-02

CONDITIONS: Phenylketonuria
Keywords: phenylketonuria ,l-carnitine, brain-derived neurotrophic factor
MeSH Terms: conditions — Phenylketonurias | interventions — Carnitine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 88 patients diagnosed as case of phenylketonuria (Experimental)
  Interventions: Drug: L-carnitine
- 88 control healthy children same age and sex (No Intervention)

INTERVENTIONS:
Drug: L-carnitine — 44 patients diagnosed as a case of phenylketonuria will receive l-carnitine at a dose of 100 mg/kg/day for 1 year and then blood sample will examined for level of brain-derived neurotrophic factor levels before and after therapy and another group composed of 44 patients diagnosed as a case of phenylketonuria will not receive l-carnitine and their blood sample will examined for level of brain-derived neurotrophic factor levels treated and untreated patients will compared with healthy children and infants has same age and sex .
  Arms: 88 patients diagnosed as case of phenylketonuria

SUMMARY:
Effect of L-carnitine supplementation on phenylalanine and brain-derived neurotrophic factor levels in infants and children with phenylketonuria

L-carnitine is mainly obtained from foods such as red meat and milk that are limited for PKU patients due to dietary protein restriction. So, L-carnitine deficiency has been described in phenylketonuric patients

The aim of this study is to :

1. Compare level of Brain-derived neurotrophic factor in infants and children with phenylketonuria and healthy infants and children.
2. Compare level of phenylalanine and Brain-derived neurotrophic factor before and after L-carnitine supplementation in phenylketonuric patients.
3. Assess Intelligence quotient test before and after L-carnitine supplementation in phenylketonuric patients

DETAILED DESCRIPTION:
Subjects And Methods :

* Type of the study: Two phases:

  1- Cross sectional comparative study ( PKU versus non PKU infants and children).

  2- Open label Randomized controlled clinical trial for PKU patients only.
* Study locality: This study will be conducted at Genetics and Metabolic Outpatient Clinic of Mansoura University Children's Hospital(MUCH).
* Study duration : assumed to conduct the research over two years.
* Inclusion criteria:

  1-Male and female PKU patients diagnosed and following up at Genetics and Metabolic Outpatient Clinic.

  2- Age from one month up to 18 years.
* Exclusion criteria:

  1. Any patient with other metabolic, genetic or neurological diseases.
  2. Patients who and/or their guardians refused to sign the consent. • Study subjects:

  1- Intervention group: Forty four patients will treated with L-carnitine at a dose of 100 mg/kg/dose for one year beside their traditional treatment.

  2- Control PKU group: Forty four patients will not receive L-carnitine supplementation beside their traditional treatment.

  3- Control healthy group: Eighty eight healthy infant and child with matched age and sex.
* Sample size:

  * All PKU pediatric patients attending to the mentioned clinic on regular follow up will be included in the study ,They are at least 88 case.
  * They will be randomized into intervention group and PKU control group(44 patients in each group).
  * An equal number of completely healthy infants and children not presented with any metabolic or genetic disorders attending to Mansoura University Children Hospital outpatient clinics will be included in the healthy control group.

    * Randomaization:

Block randomization with block size of 4 and 22 blocks using opaque sealed envelop.

Investigations:

1. Laboratory investigation:

   - Serum phenylalanine level.

   - Plasma/serum level of Brain-derived neurotrophic factor (BDNF).

   - Samples will be drawn twice for the intervention group and PKU control group basal and after one year from L- carnitine supplementation to the intervention group ,and will be drawn once for the healthy control group .

   b - Psychological assessment:

   - Stanford binet intelligence test (version 5) for children more than 3 years old.

   - Vineland adaptive behavior scale for infants and children less than 3 years.

   samples collection: For this study 5 ml whole blood samples will be collected from patients diagnosed with Phenylketonuria at Genetics and Metabolic outpatients clinic of MUCH. The plasma/serum will be separated and utilized to measure levels of phenylalanine and BDNF level by ELISA in clinical pathology lab of faculty of medicine - Mansoura university.

   Statistical analysis:

   The collected data will be coded, processed and analyzed using SPSS program (Version 29) .

   The appropriate statistical tests will be used when needed. P values less than 0.05 (5%) will be considered to be statically significant.

   Ethical consideration:
   * Study protocol will be submitted for approval by IRB.
   * Informed written consent will be obtained from each participant sharing in the study.
   * Confidentiality and personal privacy will be respected in all levels of the study. Collected data will not be used for any other purpose

ELIGIBILITY:
Inclusion Criteria:

1. Male and female PKU patients diagnosed and following up at Genetics and Metabolic Outpatient Clinic.
2. Age from one month up to 18 years

Exclusion Criteria:

1. Any patient with other metabolic, genetic or neurological diseases.
2. Patients who and/or their guardians refused to sign the consent

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 176 (Actual)
Dates: Start 2025-02-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
improve brain-derived neurotrophic factor levels | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University, Al Mansurah, Egypt